CLINICAL TRIAL: NCT02624011
Title: Influence of Increased Sedentary Time on Long-term Rates of Skeletal Muscle Protein Synthesis in Young Adults
Brief Title: Influence of Sedentary Time on Skeletal Muscle Protein Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ERN_15-1238
Record Dates: First submitted 2015-12-02; First posted 2015-12-08 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Physical inactivity (Experimental): Study arm consisting of 7 days of habitual physical activity followed by 7 days of step reduction and exercise cessation.
  Interventions: Behavioral: 7 days of habitual physical activity followed by 7 days of reduced physical activity

INTERVENTIONS:
Behavioral: 7 days of habitual physical activity followed by 7 days of reduced physical activity — Young, active participants will undergo a 7 day period of habitual physical activity followed by a 7 day period of step reduction and exercise cessation.

SUMMARY:
This study will investigate the influence of increased sedentary time on long-term measures of muscle protein synthesis and metabolic health. The investigators will test the hypothesis that increased time spent in sedentary behaviours will lead to a reduction in long-term measures of muscle protein synthesis and compromised metabolic health.

DETAILED DESCRIPTION:
Sarcopenia, the loss of muscle mass with age, is thought to be accelerated by an inactive, sedentary lifestyle. Increased sedentary time has consistently been associated with lower muscle mass and compromised metabolic health. However, there is currently a lack of direct evidence to support these associations.

Therefore, this study will investigate whether increased sedentary time (reduced step count and exercise cessation) directly influences long-term measures of muscle protein synthesis and metabolic health in young, active adults. Following a 7 day period of normal habitual physical activity, participants will undertake a 7 day period of step reduction and exercise cessation. It is hypothesised that 7 days of increased sedentary time will result in a reduction in long-term rates of muscle protein synthesis and a worsening of metabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (18.5-29.99 kg/m2)
* Active - defined as: ≥ 7000 steps per day (assessed during screening) and taking part in regular exercise (defined as participation in ≥ 3 sessions of aerobic and/or resistance exercise type sessions a week for ≥ 6 months prior to recruitment)
* Good general health

Exclusion Criteria:

* Lidocaine allergy
* Hypertension (≥140/90 mmHg)
* Current participation in another clinical study
* Previous participation in this study
* Bleeding disorder/s
* Current or recent smoker
* Past history of substance abuse and/or taking prescription or non-prescription medication (e.g., beta-blockers, insulin or thyroxine) or supplements that may influence normal metabolic responses.
* Participants who have previously (within 5 years of the present study) had 4 or more muscle biopsies obtained from the thigh quadriceps region will be ineligible.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis (FSR %/day) | 0-14 days
  Long-term muscle protein synthesis (FSR %/day) will be determined using deuterium oxide (D2O) to compare muscle protein synthesis rates over the first 7 day period and the second 7 day period.

SECONDARY OUTCOMES:
Rate of fat oxidation at rest (g/min) | For 20 minutes at day 7 and day 14
  Whole body oxygen consumption (VO2, L/min) and carbon dioxide production (VCO2, L/min) at rest will be measured using indirect calorimetry to calculate the rate of fat oxidation at rest (g/min).
Rate of fat oxidation during an oral glucose tolerance test (g/min) | At 0, 30, 60, 90 and 120min of the oral glucose tolerance test at day 7 and day 14
  Whole body oxygen consumption (VO2, L/min) and carbon dioxide production (VCO2, L/min) following an oral glucose drink will be measured using indirect calorimetry to calculate the rate of fat oxidation during an oral glucose tolerance test (g/min).
Rate of carbohydrate oxidation at rest (g/min) | For 20 minutes at day 7 and day 14
  Whole body oxygen consumption (VO2, L/min) and carbon dioxide production (VCO2, L/min) at rest will be measured using indirect calorimetry to calculate the rate of carbohydrate oxidation at rest (g/min).
Rate of carbohydrate oxidation during an oral glucose tolerance test (g/min) | At 0, 30, 60, 90 and 120min of the oral glucose tolerance test at day 7 and day 14
  Whole body oxygen consumption (VO2, L/min) and carbon dioxide production (VCO2, L/min) following an oral glucose drink will be measured using indirect calorimetry to calculate the rate of carbohydrate oxidation during an oral glucose tolerance test (g/min).
Blood glucose concentration | At 0, 30, 60, 90 and 120min of the oral glucose tolerance test at day 7 and day 14
  Blood glucose concentration will be assessed in blood samples taken during the oral glucose tolerance test.
Blood insulin concentration | At 0, 30, 60, 90 and 120min of the oral glucose tolerance test at day 7 and day 14
  Blood insulin concentration will be assessed in blood samples taken during the oral glucose tolerance test.
Blood fatty acid concentration | At 0, 30, 60, 90 and 120min of the oral glucose tolerance test at day 7 and day 14
  Blood fatty acid concentration will be assessed in blood samples taken during the oral glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon J Shad, BSc, Principal Investigator — University of Birmingham
Locations (1):
- School of Sport Exercise and Rehabilitation Sciences, University of Birmingham, Birmingham, United Kingdom